CLINICAL TRIAL: NCT02091037
Title: Staphylococcus Aureus Colonization in Atopic Dermatitis
Brief Title: S. Aureus Colonization in Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Sponsor
Other Study IDs: AAAI5956
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Bacterial colonization
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Skin culture specimens are retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to characterize the bacterial strains that colonize children with atopic dermatitis.

The investigators hypothesize that rectal cultures will be more sensitive than anterior nares cultures for detecting S. aureus colonization, and that strains of S. aureus colonizing patients with atopic dermatitis will be resistant to commonly used topical antibiotic ointments.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory skin disease characterized by pruritis and eczematous lesions with a worldwide prevalence of 15-20%. The burden of disease is highest in the most developed nations and predominantly affects children, with 50% of cases arising in the first year of life, and most others arising in the first 5 years. There is a well-known increased susceptibility to skin infection with S. aureus in patients with AD, and such infections are associated with clinical deterioration. While it is routine to evaluate for S. aureus colonization in the anterior nares, there is recent evidence suggesting that rectal colonization may be more significant. The significance of colonization site has not been evaluated in the AD population.

Additionally, while topical antibiotics are a mainstay of treatment in AD, there is no routine data on the resistance to these agents.

Our aim is to characterize the S. aureus colonization patterns in children with AD, including site of colonization and antibiotic resistance. We will analyze routinely-collected skin culture specimens from children with AD seen at our center and determine antibiotic susceptibility profiles. The significance of colonization site will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a diagnosis of atopic dermatitis seen by the Columbia University Medical Center department of dermatology
* subjects ages 0 to 18 years

Exclusion Criteria:

* those patients in which a definitive diagnosis of AD cannot be made
* subjects over the age of 18 years old
* subjects with evidence of acute systemic illness
* subjects currently taking systemic antibiotics
* subjects with viral or fungal skin infection
* any individual who declines participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the pediatric dermatology faculty practices and resident clinics at CUMC as well as from the units of the Morgan Stanley Children's Hospital of New York. As per CUMC policy, the investigators will not directly approach potential subjects until the subject's physician has ascertained and documented that their patient is willing to discuss the research with the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Difference in rectal and nasal S. aureus colonization rates in a population of children with atopic dermatitis | Up to 3 years

SECONDARY OUTCOMES:
Rates of resistance to commonly used topical antibiotic ointments in strains of S. aureus that colonize a population of children with atopic dermatitis | Up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine T Lauren, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center / Department of Dermatology, New York, New York, United States